CLINICAL TRIAL: NCT06240325
Title: A Sleep Promotion Program for Depressed Adolescents in Pediatric Primary Care
Brief Title: Sleep Promotion Program Primary Care
Acronym: SPP PC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jessica Levenson, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY23010211 (RCT); R34MH132724 (NIH)
Record Dates: First submitted 2024-01-24; First posted 2024-02-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Sleep; Sleep Disturbance; Insufficient Sleep
MeSH Terms: conditions — Parasomnias; Sleep Deprivation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Promotion Program (Experimental): Participants will receive the Sleep Promotion Program (SPP), consisting of 2 individual sessions with a clinician via telehealth (or in-person if desired), about 2 weeks apart, and web-based intervention components.
  Interventions: Behavioral: SPP
- Sleep Psychoeducation (Active Comparator): Participants will receive Sleep Psychoeducation (SPE), a 20-minute discussion with a clinician via telehealth (or in person).
  Interventions: Behavioral: Sleep Psychoeducation

INTERVENTIONS:
Behavioral: SPP — SPP prioritizes increasing sleep duration and regularizing sleep-wake timing. The provider and youth review the youth's sleep pattern, based on sleep diary data collected before and during the program and actigraphy data collected at baseline. They discuss benefits to the current sleep pattern, reasons for changing sleep, and they create an action plan. Psychoeducation about healthy sleep is offered via a handout developed by our group. Youth and provider jointly select SPP strategies relevant to the contributors to poor sleep for each youth (e.g., time management, limiting weekend oversleep). In the second session they review progress and adjust the plan. Parents participate for part of each session to learn about their child's sleep and to discuss ways they can support their child to make the planned changes.
  Arms: Sleep Promotion Program
Behavioral: Sleep Psychoeducation — Using the pamphlet also used in SPP, SPE will present sleep hygiene practices commonly included in sleep education programs and endorsed by national health organizations.
  Arms: Sleep Psychoeducation

SUMMARY:
Investigators developed a brief, scalable, behavioral Sleep Promotion Program (SPP) for adolescents with short sleep duration and sleep-wake irregularity, which relies on two individual sessions and smart phone technology to deliver evidence-based strategies. This R34 will test the feasibility and initial effectiveness of the SPP program and provider training via pilot randomized controlled trial (RCT, n=50) comparing SPP to Sleep Psychoeducation, a brief session on healthy sleep habits. Participants will be adolescents (12-18 years) with short sleep duration, sleep-wake irregularity, and depression.

ELIGIBILITY:
Inclusion Criteria:

Youth:

* Able and willing to provide informed assent (with consent from parent/guardian)
* Ages 12-18
* Currently a patient at Kids Plus Pediatrics
* Currently depressed
* Report short sleep duration (<7 hours on school nights) and/or weekday-weekend sleep timing difference of >=2 hours

Parents:

Parents must be age 18 or older and the parent/guardian of an enrolled youth participant and must have at least 10 hours face-to-face interaction with the youth participant per week.

Exclusion Criteria:

Youth:

* Significant or unstable medical conditions
* Diagnosis of sleep apnea, narcolepsy, restless leg syndrome, nightmare disorder, or periodic limb movement disorder
* Diagnosis of PTSD, bipolar disorder, a psychotic disorder, or substance use disorder
* Currently engaged in cognitive and/or behavioral therapy that aims to improve sleep
* Changes in medications in the month prior to screening
* Active suicidality requiring immediate treatment
* Unable or unwilling to comply with study procedures
* Have any physical or mental condition that would preclude study participation.

Parents will be excluded if they:

* Express active suicidality that requires immediate treatment;
* Have any physical or mental condition that would preclude study participation; OR
* Are unable or unwilling to comply with study procedures.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure | Post-Intervention (~8 weeks)
  The Feasibility of Intervention Measure (FIM) is a 4-item measure that assesses the feasibility of the intervention, each item is scored on a 1-5 likert scale (completely disagree to completely agree). Items can be evaluated individually or a scale can be created by averaging responses. Scale values range from 1-5.
Acceptability of Intervention Measure | Post-Intervention (~8 weeks)
  The Acceptability of Intervention Measure (AIM) is a 4-item measure that assesses the acceptability of the intervention, each item is scored on a 1-5 likert scale (completely disagree to completely agree). Items can be evaluated individually or a scale can be created by averaging responses. Scale values range from 1-5.
Intervention Appropriateness Measure | Post-Intervention (~8 weeks)
  The Intervention Appropriateness Measure (IAM) is a 4-item measure that assesses the appropriateness of the intervention, each item is scored on a 1-5 likert scale (completely disagree to completely agree). Items can be evaluated individually or a scale can be created by averaging responses. Scale values range from 1-5.
Clinical Global Impressions Scale - Improvement | Post-Intervention (~8 weeks)
  This is a clinician rating of improvement in sleep and psychopathology. Clinicians rate domains of sleep health, psychiatric symptoms, and overall health on a range from 1 very much improved) to 7 (very much worse). A score of 0 indicates no assessment. Scores for each domain are reported individually.
Patient Health Questionnaire - 9 - M | Change Screening to Post-Intervention (~10 weeks)
  This is a self-report measure of depressive symptoms. It consists of 9 items rated 0 (not at all) to 3 (nearly every day) over the past 2 weeks. Scores on those 9 items are summed to create a total score (0-27, higher score indicates greater depression).

SECONDARY OUTCOMES:
Pediatric Sleep Survey Sleep Knowledge (SK) | Training Start to End of Study Involvement (Up to 2.5 years)
  This is a provider self-report of knowledge about sleep. The sleep knowledge domain has 21 items that assess provider knowledge or sleep. The response options are true, false, or don't know. The number or percentage of correctly scored items is reported.
SPP Therapy Rating Scale | Completed at each SPP Session (2 and 4 weeks after baseline)
  This is a form completed by an independent rater who will review session recordings and rate them for fidelity. The scale has 5 items rated no (0) or yes (1), and 24 items rated 0 (not discussed/delivered) to 3 (excellent use of the skill). Items can be reported individually or can be summed to obtain a total score. Scale score range is 0 to 77
Sleep Diary Sleep Duration | Baseline to Post-Intervention (~8 weeks)
  This is a youth daily self-report of sleep, from which will be extracted sleep duration, reported in hours and minutes.
Sleep Diary Sleep-Wake Regularity | Baseline to Post-Intervention (~8 weeks)
  This is a youth daily self-report of sleep, from which will be extracted sleep regularity, reported as difference in sleep-wake timing between weekdays and weekends.
Quick Inventory of Depressive Symptoms - Adolescent (17 item) - Self-Report (QIDS-A17-SR) | Baseline to Post-Intervention (~8 weeks)
  This is a secondary measure of youth depression, completed by self-report, with 17 items rated on a 0 to 3 likert scale. The total score is made by summing some of the items with a total score range of 0-27.
Pediatric Sleep Survey PC | Training Start to End of Study Involvement (up to 2.5 years)
  This is a provider self-report of their comfort and capacity delivering the SPP intervention. The comfort and capacity domain asks about provider comfort delivering 14 behavioral sleep strategies, with responses on a likert scale from not at all comfortable to very comfortable. Responses can be reported individually, as well as a percentage of strategies that providers stated they were somewhat or very comfortable providing.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica C Levenson, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the National Institute of Mental Health (NIMH) Data Archive Data Use Certification, investigators will share data collected as part of this proposal with outside investigators. To access data from this study, outside investigators will be asked to submit a proposal that incudes project aims and hypotheses, variables and analytic approach, and rationale for the proposed analysis. The proposal would also include information on how and where the data will be used, investigators' qualifications, timeframe in which data will be analyzed/submitted/published, source of financial support, and conflict of interest statement. They will be asked to sign a data sharing agreement and confidentiality statement prior to the sharing of this data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All quantitative data will be cleaned and available for addressing other research questions (those not described in funded/pending grants) within one year of the completion of the study.
Access Criteria: Access to data will be provided to those meeting our pre-requesites through the National Database for Clinical Trials (NDCT) Data Access Committee (DAC). Only Investigators and Institutions who have met security measures and have submitted a Data Use Certification co-signed by the PI and the designated Institutional Official at the NIH-recognized sponsoring institution with a current Federal Wide Assurance will be given access. Outside Investigators will be asked to acknowledge the grant that supported the data collection and management in all publications and presentations.